CLINICAL TRIAL: NCT05752149
Title: The STELLAR Trial: Fluorescence-guided Surgery in Laryngeal- and Hypopharyngeal Cancer: a Feasibility Trial
Brief Title: Fluorescence-guided Surgery in Laryngeal- and Hypopharyngeal Cancer: a Feasibility Trial
Acronym: STELLAR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Stijn Keereweer, Otorhinolaryngologist, Head and Neck Surgeon, MD, PhD, Erasmus Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL74742.078.21
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Squamous Cell Carcinoma of the Larynx; Squamous Cell Carcinoma of the Hypopharynx
Keywords: Tumour specific fluorescence imaging
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The pathologist will be initially blinded during intraoperative assessment of the fresh surgical specimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 0.05 mg/kg cRGD-ZW800-1 (Experimental): n=3. Injection of 0.05 mg/kg cRGD-ZW800-1, within 2 hours before imaging/surgery
  Interventions: Drug: CRGD-ZW800-1
- 0.025 mg/kg cRGD-ZW800-1 (Experimental): n=3. Injection of 0.025 mg/kg cRGD-ZW800-1, within 2 hours before imaging/surgery
  Interventions: Drug: CRGD-ZW800-1
- 0.01 mg/kg cRGD-ZW800-1 (Experimental): n=3. Injection of 0.01 mg/kg cRGD-ZW800-1, within 2 hours before imaging/surgery.
  Interventions: Drug: CRGD-ZW800-1
- Expansion Cohort (Experimental): n=18: expansion cohort will be added to the group of patients that had received the selected dose in WP-I.
  Interventions: Drug: CRGD-ZW800-1

INTERVENTIONS:
Drug: CRGD-ZW800-1 — Intravenous administration of study drug at lesat 2h prior to surgery

SUMMARY:
This is an open-label, single-dose, prospective clinical trial. The study comprises 2 work packages. The main objective of work package I (WP-1) is to assess feasibility of Fluorescence imaing (FLI) during total laryngectomy (TLE) and to assess the optimal dose of the cRGD-ZW800-1. Work package II (WP-II) is designed to assess whether FLI can detect and decrease tumor positive margins after a TLE.

DETAILED DESCRIPTION:
This is a two staged clinical trial to investigate intraoperative fluorescence imaging in patientsundergoing TLE. WP-I is a dose finding study in which 2 doses will be tested with a possibility of a third dosing group. Every dosing cohort comprises 3 patients. After WP-I, an interim analysis will be performed to decide the optimal dose.

The optimal dose will be based on the TBR and the performance in detecting the most close margin (i.e. 'the sentinel margin'). A TBR of at least 1.5 is required for the optimal dose. If a positive margin is missed with fluorescence imaging, the concerned dose will be defined as suboptimal.

WP-II is an extension cohort of the optimal dose cohort selected in WP-I. WP-II will comprise of 18 patients.

The endpoints for WP-II are:

* the rate of tumor free resection margins based on the current golden standard;
* Sensitivity, specificity and positive predictive value of FLI;
* The intraoperative change in surgical management based on FLI;
* FLI of excised cervical lymph nodes;
* Influence of previous radiotherapy on the FLI performance;
* Adverse events and toxicity after intravenous injection with cRGD-ZW800-1;

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven squamous cell Laryngeal and hypopharyngeal cancer, eligible for surgical resection of the tumor by TLE;
* ≥ 18 years of age;
* Written informed consent must be obtained;
* Sufficient knowledge of the Dutch language to understand the informed consent form;

Exclusion Criteria:

* History of a clinically significant allergy or anaphylactic reactions to any of the components of the agent;
* Other synchronous biopsy proven malignancies currently active, except for adequately treated in situ carcinoma of cervix and basal, squamous cell skin carcinoma, or other head- and neck squamous cell cancer;
* Patients pregnant or breastfeeding;
* Patients with renal insufficiency (defined as eGFR < 60);
* Patients with previous kidney transplantation or a solitary functioning kidney;
* Patients using medications that may significantly impair renal function (i.e. NSAIDs, particularly COX-2 inhibitors), that cannot be paused during the course of the study;
* Patients with ASA classification of 4 or higher;
* Patients with measured QTc of 500 ms or higher at screening;
* Patients with laboratory abnormalities defined as:

  * Aspartate AminoTransferase, Alanine AminoTransferase, Gamma Glutamyl Transferase) or Alkaline Phosphatase levels above 5 times the ULN or;
  * Total bilirubin above 3 times the ULN or;
  * Platelet count below 100 x 109/L or;
  * Hemoglobin below 4 mmol/L (females) or below 5 mmol/l (males).
* Immuno-compromised patients who do not have the ability to respond normally to an infection due to an impaired or weakened immune system, caused by either a preexisting disease or concomitant medications;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
WP-I: the optimal dose of cRGD-ZW800-1 for FLI of laryngeal and hypopharyngeal cancer | Up to 48 hours after administration (Depending on pathology grossing)
  Based on the tumor-to-background ratio (TBR) on breadloaves. Higher TBRs indicate a better outcome
WP-II: the rate of clear tumor resection margins | Through histopathology, up to max 4 weeks post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Uponr reasonable reasonable request

REFERENCES:
- See also: Guided by Light trial — https://clinicaltrials.gov/ct2/show/NCT04191460?term=guided+by+light&draw=2&rank=1